CLINICAL TRIAL: NCT01422174
Title: Clinical Registry on Sudden Death Primary Prevention at Latin America (rEgiStro Clinico en America Latina de Prevencion Primaria en muErte Subita)
Brief Title: Clinical Registry on Sudden Death Primary Prevention at Latin America
Acronym: ESCAPE-ICD
Status: Withdrawn | Type: Observational
Why Stopped: Study stopped due to lost of interest.
Sponsor: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Other Study IDs: TA098
Record Dates: First submitted 2011-08-18; First posted 2011-08-23 (Estimated); Last update posted 2015-03-03 (Estimated); Status verified 2015-03

CONDITIONS: Myocardial Infarction; Sudden Death
Keywords: Primary prevention; Latin America; Sudden death; Myocardial infarction; Ejection Fraction; ICD
MeSH Terms: conditions — Myocardial Infarction; Death, Sudden

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ICD implantation: Patients that receive an ICD implantation (non randomized, by clinical decision) will enter this group
  Interventions: Procedure: Implantable Cardio Defibrillator (ICD),
- Non ICD implantation: Patients that do not receive ICD implantation (non randomized, by clinical decision); they can receive any other treatment (e.g. antiarrhythmic drugs)

INTERVENTIONS:
Procedure: Implantable Cardio Defibrillator (ICD), — Standard ICD implantation (as per clinical decision)
  Other Names: CE approved devices
  Groups: ICD implantation

SUMMARY:
INTRODUCTION: Sudden cardiac death is one of the most important reasons of death at industrialized countries. Despite its importance, nowadays Clinical Guidelines are not as extended as expected, with respect to indications for primary prevention defibrillator implantation, following MADIT II and MUSTT criteria, especially at Latin American countries.

OBJECTIVES: This Project is designed with the purpose of providing tools to help spreading primary prevention by the means of clinical evidence on real risk of death in this group of patients.

REGISTRY DESIGN:

* retrospective (at stage 1); prospective (at stage 2)
* multi-center (minimum 25-30 centres)
* international (Argentina, Brazil, Colombia, Chile, Mexico and Venezuela)
* non randomized.
* Sample size: at screening about 12.500 patients and 962 patients at treatment stage

REGISTRY DEVICES: CE marked (Conformité Européenne) single-chamber, dual-chamber or CRT (Cardiac Resynchronization Therapy) implantable cardiac defibrillator (ICD).

DETAILED DESCRIPTION:
REGISTRY STAGES 2 stages will be performed:

* Stage 1 (Screening): 12500 patients with MI and LVEF<40% will be evaluated, to know ICD implantation prevalence in such patients at Latin American countries
* Stage 2 (Treatment): after patient screening and as per clinical decision, 962 patients will be entered in group 1 and 2 (481 each, 1:1)

STEERING COMMITTEE

* Dr. Sergio Dubner. Clinica y Maternidad Suizo Argentina and De Los Arcos Sanatorio. Buenos Aires - Argentina
* Dr. William Uribe. CES CARDIOLOGIA. Medellin - Colombia

CLINICAL ASSESSMENT

• Dr Francisco Javier Alzueta Rodriguez. Hospital Clinico Universitario Virgen de la Victoria. Malaga - Spain

REGISTRY DURATION

* Patient enrollment period initiation: September 2011
* End of patient enrollment: September 2013
* End of FUs: September 2018
* Registry closure and data analyses: 4Q 2018.

REGULATORY CONSIDERATIONS As this is an observational registry, no submission to National Authorities is required.

ELIGIBILITY:
Inclusion Criteria:

* Patients that had Acute Myocardial Infarction (>40 days post-AMI) documented with the presence of Q-wave or cardiac-specific enzymatic markers of myocardial necrosis (CK-MB/troponin), occurred within 3 years previous to enrollment / after June 2008.
* Left Ventricular Ejection Fraction (LVEF) ≤40% post-revascularization (if no revascularization, measurement performed <3 months previous to patient enrollment, >40 days post-AMI and >3 months post-revascularization -if applicable-).

Exclusion Criteria:

* Patient with an implanted ICD
* <18 years old
* Pregnant or breast feeding women
* Patients that are already participating in other Investigational Study or Registry
* Non signed patient informed consent or refusal from patient's reference physician to patient participation
* Patient inability to comply with protocol (assist to scheduled follow-ups), due to: residence displacement out of center's activity area; unstable geographical situation or at very long distance from the center; unstable medical and/or psychological condition
* Cardiac transplanted (or in transplant waiting list)
* Severe Heart Failure (or other co-morbidity: cancer, renal failure, etc.)
* Life expectancy lower than 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at Latin American countries that fulfill MADIT, MADIT II and/or MUSTT criteria.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-03; Primary Completion 2015-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of patients with MADIT, MADIT II and MUST at Latin American countries | Patients that suffered from MI in the last 3 years and during the enrollment period
  Primary Outcome at Stage 1: Determine prevalence of patients with myocardial infarction and high risk of sudden death at Latin America, that fulfill inclusion criteria
  Primary Outcome at Stage 2: Compare MACE development in patients that receive ICD implantation vs patients that receive other type of treatment (non ICD)

SECONDARY OUTCOMES:
Study incidence of Arrhythmic mortality and serious arrhythmic events, evaluated through remote monitoring | 5 years (until end 2018)

CONTACTS AND LOCATIONS:
Overall Officials: Sergio J Dubner, MD, FACC, Principal Investigator — Clínica y Maternidad Suizo Argentina and De Los Arcos Sanatorio. Buenos Aires, Argentina; William Uribe, MD, Principal Investigator — CES Cardiología. Medellin, Colombia; Francisco J Alzueta Rodriguez (Study Clinical Advisor), Dr, Study Chair — Hospital Clínico Universitario Virgen de la Victoria. Málaga, Spain
Locations (1):
- Centro Privado de Cardiologia, San Miguel de Tucumán, Tucumán Province, Argentina